CLINICAL TRIAL: NCT07222644
Title: Clinical Language Evaluation With AI for Residents (CLEAR2) - A Pilot Randomized Controlled Trial
Brief Title: Clinical Language Evaluation With AI for Residents
Acronym: CLEAR2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Health Science Education Small Grants Program (Unknown)
Responsible Party: Principal Investigator, Krislynn Michelle Mueck, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-25-0920
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Patient Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational LLM-based feedback tool (Experimental)
  Interventions: Behavioral: educational LLM-based feedback tool
- Control (No Intervention)

INTERVENTIONS:
Behavioral: educational LLM-based feedback tool — Participants will have their verbal communications with standardized patients (SP) regarding 3 different scenarios recorded, transcribed, and analyzed in real-time by the large language model (LLM) and will receive feedback as suggestions and alternative scripts. These will be reviewed by residents between SP scenarios
  Arms: Educational LLM-based feedback tool

SUMMARY:
The purpose of this study is to refine and test existing enterprise-grade large language model (LLM) based on generative artificial intelligence (AI), to assess the feasibility and acceptability of LLM-based feedback, to assess the ability of LLM-based feedback to improve residents' communications,to explore the ability of standardized patients to assess residents' communication and to explore the ability of residents to self-assess their communication complexity

ELIGIBILITY:
Inclusion Criteria:

* McGovern Medical School (MMS) general surgery residents
* postgraduate year (PGY) 1-5

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-10-23 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Readability discernment as assessed by a survey | end of intervention ( 1 hour after baseline)
  This will be scored by the by Cohen's Kappa values from 1-5. Higher Cohen's kappa scores mean better outcome
Quality discernment as assessed by a survey | end of intervention ( 1 hour after baseline)
  This will be scored by the by Cohen's Kappa values from 1-5. Higher Cohen's kappa scores mean better outcome
Correctness of recommendations as assessed by a survey | end of intervention ( 1 hour after baseline)
  This will be reported on a 5 point Likert scale form 1 very incorrect to 5 very correct
Applicability of recommendations as assessed by a survey | end of intervention ( 1 hour after baseline)
  This will be reported on a 5 point Likert scale form 1 very inapplicable to 5 very applicable
Perceived readability of resident-standardized patient (SP) interactions as assessed by a survey: schooling level | end of intervention ( 1 hour after baseline)
  This will be categorically reported in the following categories:
  Elementary middle high college graduate
confidence in communication ability | end of intervention ( 1 hour after baseline)
  This is scored from 1( very unconfident) to 5 (very confident)
usefulness of the LLM | end of intervention ( 1 hour after baseline)
  This is scored from 1( very useless) to 5 (very useful)
acceptability of future use | end of intervention ( 1 hour after baseline)
  This is scored from 1( very unlikely) to 5 (very likely)

SECONDARY OUTCOMES:
Survey feedback on the LLM interface | end of intervention ( 1 hour after baseline)
  This is scored from 1( very unrealistic) to 5 (very realistic)
readability grade level of resident-SP transcripts as assessed by the Flesch-Kincaid Grade Level (FKGL) readability tool | end of intervention ( 1 hour after baseline)
  Readability of resident-SP encounter transcripts will be assessed using the Flesch-Kincaid Grade Level formula, which estimates the U.S. school grade level required to understand the text. Higher scores indicate a higher reading grade level (i.e., lower readability).
  Formula used:
  Grade level= 0.39(total words/total sentences) + 11.8 (total syllables/total words)-15.59
Quality based on Ensuring Quality Information for Patients (EQIP) score of resident-SP transcripts | end of intervention ( 1 hour after baseline)
  Percentage score based on a validated questionnaire This has 20 questions and each is scored from 1(yes), 0.5(partly), 0 (no) and question is removed if it does not apply.Scores are reported as a percentage and higher percentage score indicates better quality
Perceived readability of SP-resident interactions as assessed by a standardized survey | end of intervention ( 1 hour after baseline)
  This will be categorically reported in the following categories:
  Elementary middle high college graduate
confidence in communication ability | end of intervention ( 1 hour after baseline)
  This is scored from 1( very unconfident) to 5 (very confident)

CONTACTS AND LOCATIONS:
Overall Officials: Krislynn M Mueck, MD, MS, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No